CLINICAL TRIAL: NCT01771796
Title: Training Effects Following Resection Surgery in Patients With Lung Cancer
Acronym: EMITOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Collaborators: Hospital de Sant Pau (Other)
Responsible Party: Principal Investigator, Esther Marco Navarro, PhD, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PSM/RHB/CR/12
Record Dates: First submitted 2013-01-10; First posted 2013-01-18 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Lung Cancer
Keywords: Exercise; lung cancer; aerobic training, resistance training; respiratory muscle training
MeSH Terms: conditions — Lung Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aerobic and muscle resistance training (Experimental)
  Interventions: Behavioral: Aerobic and muscle resistance training
- Usual care group (No Intervention): All patients (intervention and usual care group) are patients with lung cancer who underwent a resection surgery.

INTERVENTIONS:
Behavioral: Aerobic and muscle resistance training — After having been allocated randomly to one of the two groups, patients of Intervention Group are encouraged to follow a training program (aerobic and endurance muscle training) during 8 weeks.
  Arms: Aerobic and muscle resistance training

SUMMARY:
The purpose of this study is to determine the potential benefits resulting from a specific training on exercise tolerance and muscle function at the medium and long-time, as well as study its effects on plasmatic mediators (sMICA, IGF-I and IGFBP-3) in patients with lung cancer following resection surgery.

DETAILED DESCRIPTION:
Surgical treatment of lung cancer (LC) leads to peripheral and respiratory muscle dysfunction (Mdys) with exercise limitation. This characteristic feature might be generated, not only for a reduced lung function, but also by deconditioning as well as respiratory and peripheral muscle dysfunction. It remains unknown the potential benefits resulting from a specific training and its effects on plasmatic mediators.

Chronic diseases are the leading cause of morbidity and mortality worldwide and is known that regular exercise has a beneficial effect on most of them. Many studies have shown the benefit of exercise in patients diagnosed with cancer, especially breast and colorectal cancer, even during active phases of specific treatment, however few studies refers to possible benefit of exercise in patients with lung cancer following surgical resection. Lung cancer is one of the most common cancers in Spain, the second in the general population and the first if we refer exclusively to the male population. Not only it is a common type of cancer, but also presents a high mortality with a survival rate at 5 years of approximately 12%. However, survival improves significantly in stage I (60-80% at 5 years) and progressively worse until stage IV (<5% at 5 years). Surgery is the treatment of choice for lung cancer in stages I and IIa. Despite the good results in terms of survival, it is not free of side effects. Depending on the extent of lung resection, it may result in functional limitations and impact on the patients' quality of life. Pulmonary lobectomy entails a significant reduction of the functional reserve: impaired lung function (FEV1 of 15%) and reduced exercise capacity (16% in the shuttle test). In contrast, in the pneumonectomy, reduced pulmonary function is disproportionately higher (FEV1 of 35%) in comparison with the exercise limitation (23%). To date we have no knowledge of studies that have specifically evaluated the effects of exercise training in these patients.

Dysfunction of the diaphragm and other respiratory muscles, prevalent in COPD (chronic obstructive pulmonary disease) patients, has important clinical implications. It associates with susceptibility to hypercapnic ventilatory failure, ineffective cough, and even higher incidence of repeated hospital admissions and mortality. Therefore, respiratory muscle weakness described in some patients justifies the need to train respiratory muscles because there is no general exercise (bicycle, legs, arms) able to induce an overload enough to achieve training effect on respiratory muscles. Since a large proportion of lung cancer patients also suffer from COPD, endurance and strength of respiratory muscles are expected to be reduced. Moreover, after lobectomy patients have some degree of peripheral muscle deconditioning, which could be linked to the loss of reserve function, but also the relative rest. Although muscle training has been successfully used to restore function in patients with various chronic diseases and frailty, there is little evidence on the beneficial effects of muscle training in patients after lung cancer surgery.

Many studies have related the insulin-like growth factor I (IGF-I) and its major regulatory proteins, Insulin-like growth factor binding protein (IGFBP-3) with various malignancies, including lung cancer. In healthy subjects with sedentary lifestyle, caloric diet leads to obesity and alterations of hormonal, metabolic and inflammatory modulate carcinogenesis. These disorders include chronic hyperinsulinemia, elevated plasma IGF-I, plasma enhanced bioavailability and increased steroid sex hormones of systemic inflammation markers. Physical exercise, in addition to its cardiovascular effects and/or muscular strength and endurance produces a response on plasmatic levels of IGF-I and IGFBP-3. This variability has been justified, in most cases, depending on type, intensity and/or duration of the exercise performed.

ELIGIBILITY:
Inclusion Criteria:

* 1) age under 80 years.
* 2) patients with lung cancer stage I or II with surgery indication.
* 3) ability to understand and accept the trial procedures and to sign an informed consent.

Exclusion Criteria:

* 1) Serious cardiovascular, neuromuscular or metabolic conditions that could interfere with the results and/or interfere with the measurements.
* 2) complementary cancer treatment pre-or post-surgery.
* 3) treatment with drugs with potential effect on muscle structure and function (steroids, anabolic steroids, thyroid hormones and immunosuppressive).
* 4) cognitive or language barriers that impede the realization of the objective of the study and / or collaboration in the exercise program.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-11; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Peak oxygen uptake (VO2peak) determined by a cardiopulmonary effort test (CPET) | 3 times a week during 8 weeks
  VO2peak is determined by a standardised incremental exercise test. Subjects are instructed to pedal in an electrically braked cycloergometer and are encouraged to continue until they are not able to sustain the target frequency (55-65 rpm). Loads are increased by 25 watts every 2 minutes. Different ventilatory, cardiovascular, metabolic and oxygenation variables are monitored throughout the test using a calibrated exercise system, a standard electrocardiograph, an automatic sphygmomanometer and a finger probe connected to the aforementioned digital recorder. Normal values published by Jones et al are used as the reference for physiological parameters, except for the maximum heart rate which was calculated from a standard equation published by Wassermann et al.

SECONDARY OUTCOMES:
Other effort parameters determined by the CPET | Before training (8-10 weeks post-surgery) and after (8-week training, 16-18 weeks post-surgery)
Peripheral muscle strength | Before training (8-10 weeks post-surgery) and after (8-week training, 16-18 weeks post-surgery)
Plasmatic levels of sMICA, IGF-I, IGFBP-3. | Before training (8-10 weeks post-surgery) and after (8-week training, 16-18 weeks post-surgery)

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - 1) Physical Medicine and Rehabilitation Dpt. Parc de Salut Mar., Barcelona, Barcelona
  - 2) Respiratory Medicine Dpt. Hospital de la Santa Creu i Sant Pau., Barcelona, Barcelona